CLINICAL TRIAL: NCT06781515
Title: Assessment of Disease Burden in Hairy Cell Leukemia
Acronym: BRAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BRAF
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Hairy Cell Leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCL, B-raf V600E-mutated patients (Other): For each patient only pheripheral and medullary blood sample and medullary biospy will be collected
  Interventions: Other: Peripheral and BM blood sample

INTERVENTIONS:
Other: Peripheral and BM blood sample — Peripheral and BM blood samples will be analyzed with the ddPCR method

SUMMARY:
Drug-free, single-center, prospective observational pilot study in hairy Cell Leukemia patients

DETAILED DESCRIPTION:
The V600E gene lesion of B-raf, specific and almost always present in patients with hairy cell leukemia, correlates with the presence of neoplastic cells, therefore of active disease. The measurement of the fractional abundance of the mutated gene, by ddPCR, could therefore constitute a method of molecular assessment of the minimal residual disease. In addition, the values of fractional abundance (FA) of the mutated allele obtained can be integrated coherently in patients' clinical context, along with their PB counts and BM findings.

Primary objective Verify whether the absence of mutation at the end of treatment, indicative of a state of complete molecular response to therapy, can represent a predictor of long treatment-free survival.

Secondary objectives Verify the association between the absence of mutation and the duration of response in patients who do not need treatment for at least 5 years after only one treatment with purine analogues (cladribine and pentostatin) and judged in CR according to current criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of HCL patients:

   1. newly diagnosed and candidates for first-line cytoreductive treatment with analogues purines or
   2. in relapse after a previous line of treatment, with indication for rescue therapy (repetition of a purine analogue; use of targeted or innovative drugs), except splenectomy or
   3. in CR for at least 5 years after a first line of treatment, in the absence of clinical alterations indicative of a state of hematological relapse, or in any case in the absence of an indication for a new line of cytoreductive therapy (time-to-next treatment exceeding 5 years).
2. Age ≥ 18 years at enrollment
3. Signature of written informed consent

Exclusion Criteria:

1. Concomitant second malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | through study completion, an average of 4 years
  Progression Free Survival (PFS)
Time to next treatment | through study completion, an average of 4 years
  Time to next treatment
Correlation between the share of mutated allele (fractional abundance) with the response to the treatment.Correlation between the share of mutated allele (fractional abundance) with the response to the treatment. | through study completion, an average of 4 years
  Correlation between the share of mutated allele (fractional abundance) with the response

SECONDARY OUTCOMES:
mutational pattern of B-raf i | through study completion, an average of 4 years
  Evaluation of the mutational pattern of B-raf in patients with HCL in long hematological response

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No